CLINICAL TRIAL: NCT01518699
Title: A Randomized, Double-Blind, Placebo- and Active-Controlled Study to Evaluate the Effect of Ha44 Gel on the ECG in Healthy Adult Subjects
Brief Title: Study to Evaluate the Effect of Ha44 Gel on the Electrocardiogram in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ha02-005
Record Dates: First submitted 2012-01-17; First posted 2012-01-26 (Estimated); Results first posted 2021-07-09 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Pediculosis
MeSH Terms: conditions — Lice Infestations | interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-dummy technique was used to mask the treatments. The test product is a gel and the positive control is a tablet. The active test product was administered with placebo positive control, while the active positive control was administered with placebo test product. The placebo group received both placebos.
Oversight: Data Monitoring Committee: No

ARMS (3):
- HA44 Abametapir Lotion (Experimental): Study drug plus positive-control placebo.
  Interventions: Drug: Ha44; Drug: Moxifloxacin Placebo
- Placebo (Placebo Comparator): Placebo plus positive-control placebo.
  Interventions: Drug: Ha44 Placebo; Drug: Moxifloxacin Placebo
- Moxifloxacin (Active Comparator): Placebo plus positive control
  Interventions: Drug: Ha44 Placebo; Drug: Moxifloxacin

INTERVENTIONS:
Drug: Ha44 — Abametapir Lotion 0.74%
  Other Names: Abametapir Lotion
  Arms: HA44 Abametapir Lotion
Drug: Ha44 Placebo — Ha44 Vehicle Gel without Abametapir
  Other Names: Abametapir Placebo
  Arms: Moxifloxacin; Placebo
Drug: Moxifloxacin Placebo — Moxifloxacin Placebo
  Arms: HA44 Abametapir Lotion; Placebo
Drug: Moxifloxacin — Moxifloxacin 400mg
  Other Names: Moxifloxacin Active
  Arms: Moxifloxacin

SUMMARY:
The purpose of this study is to Evaluate the Effect of Ha44 Gel on the Electrocardiogram in Healthy Volunteers.

DETAILED DESCRIPTION:
This study was a randomized, double-blind, placebo- and active-controlled, crossover study that evaluated the potential of Abametapir to prolong cardiac repolarization in healthy adult subjects (total of 57 subjects).

ELIGIBILITY:
Inclusion Criteria:

* healthy male or female subject, 18 to 50 years of age, inclusive, at least 45 kg and has a body mass index (BMI) of 18 to 33 kg/m2,
* Female subjects of childbearing potential must not be pregnant and not lactating or prepared to practice highly effective birth control methods
* The subject has normal 12-lead ECG results or, if abnormal, the abnormality is not clinically significant (as determined by the investigator).

Exclusion Criteria:

* has evidence of cardiac conduction abnormalities
* history of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmia or torsade de pointes, structural heart disease, or family history of Long QT syndrome (suggested by sudden death of a close relative due to cardiac causes at a young age
* potassium, calcium, or magnesium levels that are below the clinical laboratory's lower limit of normal
* laboratory test results at Screening are >2 x the upper limit of normal (ULN) for alanine aminotransferase (ALT) or aspartate aminotransferase (AST), >1.5 x ULN for bilirubin, or >1.5 x ULN for creatinine
* history or evidence of any clinically significant (as determined by the investigator) cardiovascular, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, and/or other major disease or malignancy (excluding non-melanoma skin cancer)
* febrile illness or symptomatic viral, bacterial (including upper respiratory infection), or fungal (non-cutaneous) infection within 1 week before clinic admission
* supine mean systolic blood pressure <90 or >140 mmHg and a mean diastolic blood pressure <50 or >90 mmHg
* positive for HIV or hepatitis C antibody or hepatitis B antigen (HBsAg)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2012-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert Dietz, MD, Principal Investigator — Spaulding Clinical
Locations (1):
- Spaulding Clinical, West Bend, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fifty seven (57) subjects were enrolled into the study. Of them 53 completed all 3 periods of the study.
Pre-assignment Details: The subjects were divided into 6 intervention arms with sequences ABC, ACB, BAC, BCA, CAB and CBA, where A is HA 44 (Abametapir) gel + Moxifloxacin placebo; B is HA 44 placebo + Moxifloxacin placebo and C is Moxifloxacin 400 mg tablet + HA 44 placebo.
Groups:
- Treatment Sequence ABC: The subjects received sequence ABC in the three periods with a 4 day washout in between two periods. In each treatment period subjects received a single dose of the treatment as follows:
  In period 1 they received HA 44 gel + Moxifloxacin placebo tablet, followed by a 4 day washout period.
  In period 2 they received HA 44 placebo + Moxifloxacin placebo, followed by a 4 day washout period.
  in period 3 they received Moxifloxacin 400 mg tablet + HA 44 placebo.
- Treatment Sequence ACB: The subjects received sequence ACB in the three periods with a 4 day washout in between two periods. In each treatment period subjects received a single dose of the treatment as follows:
  In period 1 they received HA 44 gel + Moxifloxacin placebo tablet, followed by a 4 day washout period.
  In period 2 they received Moxifloxacin 400 mg tablet + HA 44 placebo, followed by a 4 day washout period.
  In period 3 they received HA 44 placebo + Moxifloxacin placebo.
- Treatment Sequence BAC: The subjects received sequence BAC in the three periods with a 4 day washout in between two periods. In each treatment period subjects received a single dose of the treatment as follows:
  In period 1 they received HA 44 placebo + Moxifloxacin placebo, followed by a 4 day washout period.
  In period 2 they received HA 44 gel + Moxifloxacin placebo tablet, followed by a 4 day washout period.
  In period 3 they received Moxifloxacin 400 mg tablet + HA 44 placebo.
- Treatment Sequence BCA: The subjects received sequence BCA in the three periods with a 4 day washout in between two periods. In each treatment period subjects received a single dose of the treatment as follows:
  In period 1 they received HA 44 placebo + Moxifloxacin placebo, followed by a 4 day washout period.
  In period 2 they received Moxifloxacin 400 mg tablet + HA 44 placebo, followed by a 4 day washout period.
  In period 3 they received HA 44 gel + Moxifloxacin placebo tablet.
- Treatment Sequence CAB: The subjects received sequence CAB in the three periods with a 4 day washout in between two periods. In each treatment period subjects received a single dose of the treatment as follows:
  In period 1 they received Moxifloxacin 400 mg tablet + HA 44 placebo, followed by a 4 day washout period.
  In period 2 they received HA 44 gel + Moxifloxacin placebo tablet, followed by a 4 day washout period.
  In period 3 they received HA 44 placebo + Moxifloxacin placebo.
- Treatment Sequence CBA: The subjects received sequence CBA in the three periods with a 4 day washout in between two periods. In each treatment period subjects received a single dose of the treatment as follows:
  In period 1 they received Moxifloxacin 400 mg tablet + HA 44 placebo, followed by a 4 day washout period.
  In period 2 they received HA 44 placebo + Moxifloxacin placebo, followed by a 4 day washout period.
  In period 3 they received HA 44 gel + Moxifloxacin placebo tablet.
Period: Period 1
Arm/Group | Treatment Sequence ABC | Treatment Sequence ACB | Treatment Sequence BAC | Treatment Sequence BCA | Treatment Sequence CAB | Treatment Sequence CBA
Started | 10 | 9 | 9 | 10 | 10 | 9
Completed | 10 | 9 | 9 | 10 | 10 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Treatment Sequence ABC | Treatment Sequence ACB | Treatment Sequence BAC | Treatment Sequence BCA | Treatment Sequence CAB | Treatment Sequence CBA
Started | 10 | 9 | 9 | 10 | 10 | 9
Completed | 8 | 7 | 9 | 10 | 10 | 9
Not Completed | 2 | 2 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Treatment Sequence ABC | Treatment Sequence ACB | Treatment Sequence BAC | Treatment Sequence BCA | Treatment Sequence CAB | Treatment Sequence CBA
Started | 8 | 7 | 9 | 10 | 10 | 9
Completed | 8 | 7 | 9 | 10 | 10 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized subjects
Groups:
- Treatment Sequence ABC: The subjects received sequence ABC in the three periods with a 4 day washout in between the periods. In each treatment period, subjects received a single dose of the treatment as follows:
  In period 1 they received HA 44 gel + Moxifloxacin placebo tablet, followed by a 4 day washout period.
  In period 2 they received HA 44 placebo + Moxifloxacin placebo, followed by a 4 day washout period.
  in period 3 they received Moxifloxacin 400 mg tablet + HA 44 placebo.
- Total: Total of all reporting groups
Arm/Group | Treatment Sequence ABC | Treatment Sequence ACB | Treatment Sequence BAC | Treatment Sequence BCA | Treatment Sequence CAB | Treatment Sequence CBA | Total
Number analyzed (Participants) | 10 | 9 | 9 | 10 | 10 | 9 | 57
Age, Customized [Mean (Standard Deviation); unit: years] | 28.1 (5.47) | 28.0 (9.04) | 28.8 (7.21) | 28.2 (6.81) | 32.6 (9.70) | 33.8 (8.66) | 29.9 (7.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 4 | 7 | 5 | 6 | 31
  Male | 7 | 3 | 5 | 3 | 5 | 3 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 1 | 4 | 1 | 1 | 9
  Not Hispanic or Latino | 8 | 9 | 8 | 6 | 9 | 8 | 48
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 1 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 5 | 6 | 3 | 2 | 3 | 22
  White | 7 | 3 | 2 | 6 | 8 | 6 | 32
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 9 | 10 | 10 | 9 | 57

OUTCOME MEASURES:

1. Primary Outcome: Difference Between Active and Placebo for Time Matched Baseline Adjusted Mean QTcF
Description: The primary endpoint is the difference between the active (HA44) and placebo for time matched baseline adjusted mean QTcF = [ΔQTcF (Ha44 0.74% Gel) - ΔQTcF (placebo)] = ΔΔQTcF. This was compared with the difference between Moxifloxacin and placebo for time matched baseline adjusted mean QTcF = [ΔQTcF (Moxifloxacin) - ΔQTcF (placebo)] = ΔΔQTcF
Time Frame: 36 hours
Population: All completed subjects
Measure: Mean (Standard Deviation); unit: milliseconds
Groups:
- HA 44 Gel + Moxifloxacin Placebo; HA 44 Placebo + Moxifloxacin Placebo: The maximal difference between baseline and post treatment value in QTcF
- Moxifloxacin 400 mg Tablet +HA 44 Placebo: The maximum difference between baseline and post treatment values in QTcF
Arm/Group | HA 44 Gel + Moxifloxacin Placebo | HA 44 Placebo + Moxifloxacin Placebo | Moxifloxacin 400 mg Tablet +HA 44 Placebo
Number analyzed (Participants) | 53 | 53 | 53
milliseconds | -9.7 (10.27) | -9.2 (10.10) | 6.1 (7.64)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the time of signing informed consent until the last study assessment i.e. for 18 days.
Groups:
- Moxifloxacin: Placebo plus Moxifloxacin
Arm/Group | HA44 Abametapir Lotion | Placebo | Moxifloxacin
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/54 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/54 | 0/53
Other Adverse Events (participants affected / at risk) | 26/57 | 3/54 | 14/53
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HA44 Abametapir Lotion (N=57) | Placebo (N=54) | Moxifloxacin (N=53)
Application site erythema (Skin and subcutaneous tissue disorders) | 11 (11) | 0 (0) | 1 (1)
Application site pain (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (5)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 4 (4)
Application site pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 6 (6) | 3 (3) | 5 (5)
Dysmenorrhoea (Reproductive system and breast disorders) | 3 (3) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No